CLINICAL TRIAL: NCT07195682
Title: A Phase 1/1b Open-label, Multi-center Study of BMS-986506 in Participants With Advanced Clear Cell Renal Cell Carcinoma (ccRCC)
Brief Title: A First-in-Human Study of BMS-986506 in Participants With Advanced Clear Cell Renal Cell Carcinoma (ccRCC)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA242-0001; 2025-522543-18 (Other: EU CTR); U1111-1323-5879 (Other: WHO)
Record Dates: First submitted 2025-09-25; First posted 2025-09-29 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Renal Cell Carcinoma
Keywords: Metastatic clear cell renal cell carcinoma; Advanced clear cell renal cell carcinoma; ccRCC; Kidney cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Clear-cell metastatic renal cell carcinoma; Kidney Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BMS-986506: Part 1A (Experimental)
  Interventions: Drug: BMS-986506
- BMS-986506: Part 2A (Experimental)
  Interventions: Drug: BMS-986506
- BMS-986506: Part 2B (Experimental)
  Interventions: Drug: BMS-986506

INTERVENTIONS:
Drug: BMS-986506 — Specified dose on specified days

SUMMARY:
This is a first-in-human study of BMS-986506 in participants with advanced Clear Cell Renal Cell Carcinoma (ccRCC). The primary objective of this study is to find out if BMS-986506 is safe and can be tolerated when taken alone by participants with ccRCC.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed diagnosis of locally advanced or metastatic ccRCC.
* For part 1: Participants must have already had at least two different treatment plans in the past, including immunotherapy and a targeted therapy.
* For part 2: Participants must have had at least one standard treatment plan that included both a PD-1/L1 inhibitor and a VEGF-TKI (either together or one after the other).
* Participants must have Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.

Exclusion Criteria:

* Participants with Inability to administer and/or tolerate oral medication without chewing, breaking, crushing, or otherwise altering the product dosage form.
* For Part 2A: Participants who have received more than 3 prior systemic regimens for locally advanced or metastatic ccRCC including prior treatment with HIF2a inhibitors.
* Participants who have hypoxia as defined by a pulse oximeter reading < 92% at rest or requires intermittent or chronic supplemental oxygen.
* Participants who have received colony-stimulating factors (eg, G-CSF, GM-CSF or recombinant EPO) within 28 days prior to the first dose of study intervention.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2026-01-15 (Actual); Primary Completion 2030-05-03 (Estimated); Study Completion 2031-04-03 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | Up to approximately 2 years from first dose of BMS-986506
Number of Participants With Serious Adverse Events (SAEs) | Up to approximately 2 years from first dose of BMS-986506
Number of Participants With AEs Meeting Protocol Defined Dose-limiting Toxicity (DLT) Criteria | Up to approximately Day 28
Number of Participants With AEs Leading to Discontinuation | Up to approximately 2 years from first dose of BMS-986506
Number of Participants With AEs Leading to Deaths as Assessed by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v 5.0 | Up to approximately 2 years from first dose of BMS-986506

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of BMS-986506 | Up to approximately Day 85
Time of Maximum Observed Plasma Concentration (Tmax) of BMS-986506 | Up to approximately Day 112
Area Under the Concentration-time Curve Within a Dosing Interval (AUC-TAU) of BMS-986506 | Up to approximately Day 112
Objective Response Rate (ORR) as Assessed by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) | Up to approximately 3 years from first dose of BMS-986506
Disease Control Rate (DCR) as Assessed by RECIST v1.1 | Up to approximately 3 years from first dose of BMS-986506
Duration of Response (DOR) as Assessed by RECIST v1.1 | Up to approximately 3 years from first dose of BMS-986506
Time to Response (TTR) as Assessed by RECIST v1.1 | Up to approximately 3 years from first dose of BMS-986506

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (9):
- United States (5):
  - Local Institution - 0006, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Local Institution - 0002, Philadelphia, Pennsylvania
  - SCRI Oncology Partners, Nashville, Tennessee
  - START San Antonio, San Antonio, Texas
- Local Institution - 0021, Calgary, Alberta, Canada
- Local Institution - 0008, Villejuif, Val-de-Marne, France
- Spain (2):
  - Local Institution - 0015, Córdoba, Andalusia
  - Local Institution - 0018, Barcelona, Barcelona [Barcelona]

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT07195682.html